CLINICAL TRIAL: NCT03261596
Title: Efficacy and Safety of a Single-dose Regimen and a Multi-dose Regimen of Mebendazole Against Hookworm Infections in Children and Adolescents in Ghana: a Randomized Controlled Trial
Brief Title: Mebendazole Study Against Hookworm Infections in Children and Adolescents in Ghana
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: In light of new evidence, the decision was made by the sponsor to not proceed.
Sponsor: PATH (Other)
Collaborators: Yale University (Other); Noguchi Memorial Institute for Medical Research (Other); Ghana Health Services (Other Government); HopeXchange Medical Center, Ghana (Unknown); Kintampo Health Research Centre, Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH-MBZ-PO-4 02-GHA
Record Dates: First submitted 2017-08-16; First posted 2017-08-25 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Hookworm Infections
Keywords: Soil-transmitted helminth; hookworm; hookworm infections; necator americanus; ancylostoma duodenale
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis | interventions — Mebendazole

STUDY DESIGN:
Intervention Model Description: The study will be a single site Phase 4, open-label, randomized controlled study. Subjects will be randomized 1:1 to one of two treatment allocations: 150 to receive a single dose of 500 mg mebendazole and 150 to receive a multi-dose of 100 mg mebendazole twice a day for three days.
Who Masked: Participant
Masking Description: Study drug will be maintained and dispensed to the participant by a qualified un-blinded study staff member and witnessed by another un-blinded study staff member. The blinding of laboratory staff will be maintained throughout the trial until data entry and processing are complete and the data have been verified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 mg solid tablets 2x/day for 3 days (Experimental): Assess the efficacy (Cure Rate/CR) and safety of 100 mg dose regimen of mebendazole in children aged 6 to 18 years, inclusive, infected with hookworm.
  Interventions: Drug: Mebendazole
- Single dose 500 mg solid tablets (Experimental): Assess the efficacy (Cure Rate/CR) and safety of 500 mg dose regimen of mebendazole in children aged 6 to 18 years, inclusive, infected with hookworm.
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — Participants will be randomized using a 1:1 ratio to one of the two arms. Study participants eligible for treatment will be randomly assigned to one of the two treatment arms using a computer-generated stratified block randomization code.
  Other Names: Vermox

SUMMARY:
The Ghana study will hypothesize that both the multiple dose and single dose of mebendazole will achieve effective cure rates against hookworm among children and adolescents. This study is intended to be a pilot study for a planned Phase 3 registration trial of a new drug for hookworm, tribendimidine.

DETAILED DESCRIPTION:
This study will determine the Cure Rates (CRs) of mebendazole regimens to be used as comparator drug regimens in the future pivotal trial of tribendimidine and will provide evidence of the efficacy and safety of mebendazole among children and adolescents infected with hookworm in Ghana. Children and adolescents bear a large burden of morbidity from hookworm infection, so building the evidence base for effective treatments in this population has important public health implications in Ghana and other endemic settings.

ELIGIBILITY:
Inclusion Criteria

All participants must meet all of the following inclusion criteria:

1. Male or female, aged 6 to 18 years, inclusive, at the time of randomization.
2. Written informed consent signed by at least one parent and/or legally acceptable representative (as defined by local law); and assent by participant.
3. Able and willing to be examined by a study health care provider at the beginning of the study.
4. Able and willing to provide one stool sample at the beginning (baseline) and one sample approximately three weeks after treatment (follow-up).
5. Positive for hookworm eggs in the stool (two Kato-Katz thick smear slides with more than one hookworm egg) at baseline.

Exclusion Criteria

Participants must meet none of the following exclusion criteria to be eligible for this study:

1. Presence of major systemic illnesses as assessed by a study health care provider, upon initial targeted clinical assessment.
2. Pregnancy, based on a positive urine rapid test, or breastfeeding in girls after menarche.
3. Recent use of an anthelminthic drug (within the past 4 weeks) or use of anthelminthics not provided by study staff during the study period.
4. Known allergy to mebendazole or albendazole.
5. Participation in other clinical trials during the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cure Rate (CR) against hookworm, as determined by Kato Katz. | 20 days
  To determine point estimates for the efficacy of two mebendazole regimens: (i) 100 mg solid tablets twice daily for three days, and (ii) single dose of 500 mg solid tablets in participants aged 6 to 18 years infected with hookworm. The CR will be calculated as the percentage of children and adolescents (all hookworm egg-positive at enrollment) who are egg negative 20 days after treatment. The CRs will be tabulated by mebendazole dose regimen received, along with their corresponding 95% CIs.

SECONDARY OUTCOMES:
Egg reduction rate (ERR), based on geometric mean, against hookworm | 20 days
  In a simple analysis, the study will estimate a risk ratio between CRs by using log binomial regression. Baseline characteristics will be assessed by arm to determine any imbalance between the two randomization arms. Any factor (e.g., age, sex, school, weight, height, baseline hookworm infection intensity) out of balance at baseline will be adjusted for in the analyses. Sensitivity analyses will be conducted which will consider all participants with missing endpoint data as treatment failure or all as treatment success to test whether the results (of the CR comparison) are sensitive to potential differences in loss to follow-up.
CR and ERR against Ascaris lumbricoides and Trichuris trichiura | 20 days
  Determine the ERR in the two treatment arms; EPG will be assessed by adding up the egg counts from the Kato-Katz thick smears and multiplying this number by twenty-four. The ERR will be calculated (ERR = (1-(mean egg count at follow-up/mean egg count at baseline))*100). Geometric mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. The bootstrap resampling method with 5,000 replicates will be used to calculate 95% CIs for ERRs and the difference between the ERRs. Analyses of mebendazole efficacy against concomitant STHs will proceed similarly to those conducted for hookworm.
Adverse Events | Through 20 days of follow-up
  For the safety objective, the probability of observing zero, one or more, and two or more solicited AEs among the 150 subjects in each treatment arm given a true event rate. For example, if the true rate of an AE among subjects receiving single dose mebendazole is 1% then the probability we will see 1 or more subjects with this event is 78%.

OTHER OUTCOMES:
Sensitivity of Kato-Katz and PCR for hookworm infection detection | Up to 14 weeks following Day 20
  Compare the sensitivity of Kato-Katz to quantitative polymerase chain reaction (PCR) assays among participants at day 20 of follow-up. As there is no true gold standard for hookworm diagnosis, we will consider individuals as "true" positives if they are identified as positive by PCR or Kato-Katz. This assumes no false positives for either diagnostic technique. While PCR has higher sensitivity than microscopy in general, microscopy has been noted to have high specificity. The study will therefore avoid discounting as "true" positives those who test negative by PCR but positive by microscopy and conduct an inter-method reliability study to separately compare hookworm and other STH diagnoses by PCR or the pooled microscopy in the full sample (N= 300) with the pooled (Kato-Katz or PCR positive) gold standard. Specificity cannot be calculated, as both diagnostic methods are contained within the pooled gold standard.
Prevalence of hookworm genetic resistance markers | Up to 14 weeks following Day 20
  Determine the prevalence of hookworm genetic resistance markers among participants at day 20 of follow-up. The conditional prevalence is defined as the proportion of individuals who have a disease subtype among those who test positive for the disease. All participants identified as positive for hookworm by PCR at day 20 will be considered hookworm positive.
Distribution of hookworm species among participants | Up to 14 weeks following Day 20
  Determine the distribution of hookworm species among participants at baseline. All participants identified as positive for hookworm by PCR at baseline will be considered hookworm positive. The conditional prevalence(s) will be calculated as follows, pooled and separately for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cappello, MD, Principal Investigator — Yale University; Michael Wilson, PhD, Principal Investigator — University of Ghana
Locations (1):
- Noguchi Memorial Institute for Medical Research - University of Ghana, Legon, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
The final results of this study will be published in a scientific journal and presented at scientific conferences. Any publication, lecture, and manuscripts of the findings of this study by any individual involved with the study will be governed by the procedure outlined in the Clinical Trial Agreement. Within any presentation or publication, confidentiality of individual subjects will be maintained, with identification by subject code number and initials, if applicable. A summary of study conclusions will be shared with the local community.